CLINICAL TRIAL: NCT00305812
Title: A Randomized Phase II Dose Finding Study of Revlimid™ and Melphalan in Patients With Previously Untreated Multiple Myeloma
Brief Title: Lenalidomide and Melphalan in Treating Patients With Previously Untreated Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MY11; CAN-NCIC-MY11 (Other: PDQ); CELGENE-CAN-NCIC-MY11 (Other: Celgene); CDR0000466184 (Other: PDQ)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-03

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Lenalidomide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: dexamethasone
Drug: lenalidomide
Drug: melphalan

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. It may also stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with melphalan may kill more cancer cells.

PURPOSE: This randomized phase II trial is studying the side effects and best dose of lenalidomide when given together with melphalan and to see how well they work in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the tolerability of 2 different doses of lenalidomide when administered with melphalan in patients with previously untreated multiple myeloma who are not planning to undergo future autologous stem cell transplantation.

Secondary

* Characterize the toxicity profile of lenalidomide in combination with melphalan.
* Determine tumor response in these patients after 2 and 12 courses of induction therapy with lenalidomide and melphalan and after 6 months of maintenance therapy with dexamethasone.
* Determine progression-free and overall survival of these patients.
* Determine time to dose modification and time to dose discontinuation in these patients.

Tertiary

* Examine wnt pathway inhibition in response to lenalidomide on pre- and post-treatment bone marrow and blood samples using enzyme-linked immunosorbent assay (ELISA), gene expression profiling, drosophila-based chemical genetics, and surface-enhanced laser desorption/ionization mass spectrometry (SELDI MS) proteomics.

OUTLINE: This is a multicenter, randomized, open-label, dose-finding study of lenalidomide.

Prior to randomization, 6 patients receive oral lenalidomide at a lower dose (same dose to be used in arm I) once daily on days 1-21 and oral melphalan once daily on days 1-4. Treatment repeats every 28 days for 3 courses. If no unacceptable toxicity occurs, the trial will proceed and randomization will occur.

* Induction therapy: Patients are randomized to 1 of 2 dose levels of lenalidomide.

  * Arm I: Patients receive oral lenalidomide once daily on days 1-21 and oral melphalan once daily on days 1-4.
  * Arm II: Patients receive oral lenalidomide as in arm I, but at a lower dose, and melphalan as in arm I, but at a higher dose.

Treatment in both arms repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. After 12 courses of induction therapy, patients in both arms without progressive disease proceed to maintenance therapy.

* Maintenance therapy: Patients receive oral dexamethasone once daily on days 1-4. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 92 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed multiple myeloma by one of the following:

  * Biopsy of an osteolytic lesion or soft tissue tumor composed of plasma cells
  * Bone marrow aspirate and/or biopsy demonstrating ≥ 10% plasmacytosis
  * Bone marrow < 10% plasma cells but with ≥ 1 bony lesion AND meets the M-protein criteria
* Ineligible for stem cell transplantation due to any of the following:

  * Advanced age
  * Comorbid illness
  * Patient preference
* Previously untreated disease
* Measurable (i.e., quantifiable) serum M-component of IgG, IgA, IgD, or IgE at initial diagnosis OR, if only light-chain disease is present (urine M-protein only), urinary excretion of light-chain protein (Bence Jones) ≥ 1.0 g/24 hours at initial diagnosis

  * No nonsecretory myeloma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 150,000/mm^3
* Creatinine ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST and/or ALT ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception during and for 4 weeks after completion of study treatment
* No other malignancies within the past 5 years, except adequately treated nonmelanoma skin cancer or curatively treated in situ cancer of the cervix
* No hypersensitivity to thalidomide or its components, including the development of a desquamating rash
* No other serious illness or medical condition that would preclude study participation
* No history of significant neurologic or psychiatric disorder that would preclude informed consent
* No known HIV positivity
* No pre-existing cardiovascular conditions and/or symptomatic cardiac dysfunction, including any of the following:

  * Significant cardiac event (including symptomatic heart failure or angina) within 3 months prior to randomization
  * Any cardiac disease that increases risk for ventricular arrhythmia
  * History of ventricular arrhythmia that was symptomatic or required treatment, including any of the following:

    * Multifocal premature ventricular contractions
    * Bigeminy
    * Trigeminy
    * Ventricular tachycardia/fibrillation/flutter/arrhythmia NOS

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or corticosteroids for the treatment of multiple myeloma

  * Prior corticosteroids for the treatment of hypercalcemia or spinal cord compression allowed provided maximum levels have not been reached (i.e.,< 120 mg for dexamethasone or < 792 mg for prednisone)
* Prior radiotherapy to single sites for pain control or local plasmacytoma allowed
* Prior or concurrent bisphosphonates allowed
* At least 28 days since prior investigational anticancer agents or therapy
* No concurrent corticosteroids above physiologic replacement doses
* Concurrent radiotherapy to sites of active myeloma with pain or neurologic compromise allowed
* No concurrent filgrastim (G-CSF) on day 1 of course 1
* No other concurrent anticancer therapy
* No other concurrent investigational therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-03-09 (Actual); Primary Completion 2008-06-30 (Actual); Study Completion 2008-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity within first 3 courses of treatment

SECONDARY OUTCOMES:
Toxicity
Disease response after 2 courses, 6 courses, 12 courses, and 6 months of maintenance therapy
Time to progression
Overall survival
Duration of disease-free interval
Time to dose modification
Time to dose discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Darrell White, MD, Study Chair — Nova Scotia Cancer Centre
Locations (14):
- Canada (14):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Moncton Hospital, Moncton, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Algoma District Cancer Program at Sault Area Hospital, Sault Ste. Marie, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Humber River Regional Hospital - Weston, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White DJ, Paul N, Macdonald DA, Meyer RM, Shepherd LE. Addition of lenalidomide to melphalan in the treatment of newly diagnosed multiple myeloma: the National Cancer Institute of Canada Clinical Trials Group MY.11 trial. Curr Oncol. 2007 Apr;14(2):61-5. doi: 10.3747/co.2007.107. PMID 17576467
- [Result] White DJ, Bahlis NJ, Marcellus DC, et al.: Phase II testing of lenalidomide plus melphalan for previously untreated older patients with multiple myeloma: the NCIC CTG MY.11 trial. [Abstract] Blood 112 (11): A-2767, 2008.
- [Result] White DJ, Kovacs MJ, Belch A, et al.: Phase II testing of lenalidomide plus melphalan for previously untreated older patients with multiple myeloma: toxicity data from the NCIC CTG MY.11 trial. [Abstract] Blood 110 (11): A-189, 2007.
- [Derived] White DJ, Bahlis NJ, Marcellus DC, Belch A, Stewart AK, Chen C, Kovacs MJ, Macdonald DA, Reece DE, Reiman T, Harnett E, Meyer RM, Chapman JA, Couban S. Lenalidomide plus melphalan without prednisone for previously untreated older patients with multiple myeloma: a phase II trial. Clin Lymphoma Myeloma Leuk. 2013 Feb;13(1):19-24. doi: 10.1016/j.clml.2012.08.009. Epub 2012 Nov 7. PMID 23141150